CLINICAL TRIAL: NCT07244302
Title: The Effect of Abdominal Massage Applied to Patients by Caregivers in Palliative Care Clinics on Gastrointestinal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AEŞH-EK-2025-153
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Symptoms
Keywords: Abdominal Massage; Gastrointestinal Symptoms; Palliative Care; Constipation; Caregivers
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Caregivers received training on abdominal massage and applied the massage to patients twice daily for 15 minutes between Days 2 and 7. Each session was recorded on the Abdominal Massage Application Follow-up Form.
  Interventions: Behavioral: Abdominal Massage
- Control Group (No Intervention): Patients in the control group received no additional intervention and continued to receive routine palliative care throughout the study period.

INTERVENTIONS:
Behavioral: Abdominal Massage — In the intervention group, caregivers received training on abdominal massage, and an Abdominal Massage Training Manual prepared by the researchers was provided to reinforce the education. Following the training, caregivers administered abdominal massage to the patients twice daily for 15 minutes between Days 2 and 7. The massage procedures were performed in accordance with the defined abdominal massage steps, using clockwise movements over the abdominal region, with the aim of reducing gastrointestinal symptoms.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to examine the effect of abdominal massage applied by caregivers to patients in palliative care clinics on gastrointestinal symptoms.

Hypotheses H0a: Abdominal massage applied by caregivers to patients in palliative care clinics has no effect on gastrointestinal symptoms.

H1a: Abdominal massage applied by caregivers to patients in palliative care clinics has an effect on gastrointestinal symptoms.

In this study, the effect of abdominal massage applied to patients following abdominal massage training provided to caregivers in the intervention group will be evaluated by comparing the intervention group, which receives abdominal massage, with the control group, which receives routine care.

DETAILED DESCRIPTION:
On the first day of the study, the aim, scope, and procedural steps were thoroughly explained to the patients and their caregivers in both groups, written informed consent was obtained, and baseline assessments were conducted. These assessments included the Individual Descriptive Characteristics Form, Barthel Index of Activities of Daily Living, Defecation Diary, Bristol Stool Form Scale, and the Gastrointestinal Symptom Rating Scale. Subsequently, caregivers in the intervention group received abdominal massage training, and the Abdominal Massage Training Manual prepared by the researchers was provided to support the correct application of the massage techniques.

In the intervention group, patients received abdominal massage administered by their caregivers twice daily for 15 minutes between Days 2 and 7, and each application was recorded on the Abdominal Massage Application Follow-up Form. Patients in the control group continued to receive routine care during the same period. In both groups, Defecation Diary parameters and the Bristol Stool Form Scale were evaluated daily by the researcher between Days 2 and 7.

At the end of Day 7, the Gastrointestinal Symptom Rating Scale was administered again, final assessments were completed, and the study was concluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified as constipated according to the Rome IV diagnostic criteria, as assessed by a clinical specialist.
* Patients whose hospitalization in the palliative care unit was planned for at least 7 days.
* Patients who were able to receive oral nutrition during the study period.
* Individuals aged 18 years or older.
* Patients who provided written informed consent, or whose first-degree relatives provided consent on their behalf.
* Caregivers responsible for administering the abdominal massage who provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients with known gastrointestinal diseases such as ulcerative colitis, Crohn's disease, or irritable bowel syndrome.
* Patients who had received abdominal radiotherapy within the last six weeks or who had undergone abdominal surgery within the past year.
* Patients with acute abdomen, colostomy or ileostomy, significant abdominal distension, abdominal hernia, abdominal tumors, diarrhea, or fecal impaction.
* Patients who were pregnant or suspected of being pregnant.
* Patients receiving enteral nutrition via percutaneous endoscopic gastrostomy (PEG), nasogastric tubes, or similar feeding methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-11-09 (Actual); Study Completion 2025-11-09 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Severity Assessed by the Gastrointestinal Symptom Rating Scale (GSRS) | Baseline (Day 1) to Day 7
  The primary outcome of this study is the change in gastrointestinal symptom severity assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS is a validated and widely used instrument consisting of 15 items organized into five subscales: abdominal pain, reflux, indigestion, diarrhea, and constipation. Each item is scored on a 7-point Likert scale (1 = no discomfort, 7 = very severe discomfort), with higher scores indicating more severe symptoms.
  The GSRS will be administered at baseline (Day 1) and again at the end of the study period (Day 7). The primary analysis will evaluate the change in the total GSRS score between Day 1 and Day 7 to determine the overall effect of the intervention.
  In addition to the total score, all five GSRS subscale scores will be analyzed separately to assess symptom-specific effects of abdominal massage. Between-group comparisons (intervention vs. control) will be conducted to evaluate whether caregiver-administered abdominal massage lead

SECONDARY OUTCOMES:
Change in Stool Consistency Assessed by the Bristol Stool Form Scale | Daily assessments from Day 1 (baseline) through Day 7
  Stool consistency will be assessed using the Bristol Stool Form Scale (BSFS) on Day 1 (baseline) and daily from Days 2 to 7. The BSFS classifies stool into seven types ranging from hard and lumpy (Type 1) to completely liquid (Type 7), providing an objective evaluation of stool form.
  Daily stool form will be recorded by the researcher, and changes from the baseline (Day 1) measurement across the 7-day follow-up period will be analyzed. Comparisons between the intervention and control groups will be performed to determine whether abdominal massage administered by caregivers influences stool consistency over time.
Change in Bowel Movement Characteristics Assessed by the Defecation Diary | Daily assessments from Day 1 through Day 7
  Bowel movement characteristics will be assessed daily using a structured Defecation Diary. The diary includes five parameters:
  number of bowel movements, stool amount (1-3 points), stool consistency (1-5 points), straining during defecation (1-4 points), sensation of incomplete evacuation (0-1 points).
  Two additional parameters are also recorded daily: laxative/enema use (yes/no), presence of gas/bloating (yes/no). Daily scores from Day 1 to Day 7 will be analyzed to determine changes in bowel function, and comparisons will be made between the intervention and control groups.

OTHER OUTCOMES:
Baseline Functional Independence Assessed by the Barthel Index | Day 1 (Baseline only)
  The Barthel Index will be used at baseline to assess the functional independence level of participants and to describe the initial characteristics of the study groups. This measure is not intended as an outcome variable and will not be used for pre-post comparisons.
Baseline Descriptive and Demographic Characteristics | Day 1 (Baseline only)
  Baseline descriptive characteristics will be collected using a structured Descriptive Information Form on Day 1. Variables include age, sex, medical diagnosis, duration of hospitalization, comorbidities, medication use, caregiver characteristics, and other relevant demographic or clinical factors. These data will be used solely to describe the study population and evaluate group comparability at baseline. They will not be analyzed as study outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma İ Çınar, Prof. Dr., Study Director — Gülhane Hemşirelik Fakültesi, Sağlık Bilimleri Üniversitesi
Locations (1):
- Ankara Etlik Şehir Hastanesi, Tıbbi Gözlem Kulesi Palyatif Bakım Kliniği, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a single-center academic thesis project and the collected data contain sensitive clinical information that cannot be made publicly available. Data will be used only for the purposes of this research and will not be shared with external investigators.